CLINICAL TRIAL: NCT02581995
Title: Open-label Phase-4 Study to Examine the Change of Vision-related Quality of Life in Subjects With Diabetic Macular Edema (DME) During Treatment With Intravitreal Injections of 2 mg Aflibercept According to EU Label for the First Year of Treatment
Brief Title: Investigation of the Change of Vision-related Quality of Life in Subjects Treated With Aflibercept According to EU Label for DME.
Acronym: AQUA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17850; 2014-005119-17 (EudraCT Number)
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Results first posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-09

CONDITIONS: Macular Edema
Keywords: Diabetic macular edema; Intravitreal injection
MeSH Terms: conditions — Macular Edema | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Arm 1 / Quality of Life (Experimental): Aflibercept treatment in subjects with diabetic macular edema (DME)
  Interventions: Drug: Eylea (Aflibercept, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Eylea (Aflibercept, VEGF Trap-Eye, BAY86-5321) — 2 mg aflibercept administered every 8 weeks following 5 initial monthly doses Intravitreal (IVT) injection

SUMMARY:
To evaluate the change in quality of life (NEI VFQ 25) in subjects with DME during the first year of treatment with aflibercept according to the EU Label.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or 2 diabetes mellitus
* Diagnosis of DME secondary to diabetes mellitus involving the center of the macula (defined as the area of the center subfield on OCT) in the study eye
* Decrease in vision determined to be primarily the result of DME in the study eye
* BCVA in the study eye of ETDRS letter score 73 to 24 (This corresponds to a Snellen equivalent of approximately 20/40 to 20/320.)

Exclusion Criteria:

* Pregnancy and lactation
* Mismatch with inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2015-11-19 (Actual); Primary Completion 2017-08-09 (Actual); Study Completion 2017-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (68):
- Austria (2):
  - Graz, Styria
  - Vienna
- Canada (7):
  - Halifax, Nova Scotia
  - London, Ontario
  - Mississauga, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Sherbrooke, Quebec
- Czechia (3):
  - Hradec Králové
  - Prague
  - Ústí nad Labem
- France (2):
  - Créteil
  - Marseille
- Germany (10):
  - Darmstadt, Hesse
  - Frankfurt am Main, Hesse
  - Marburg, Hesse
  - Göttingen, Lower Saxony
  - Bonn, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Ludwigshafen am Rhein, Rhineland-Palatinate
  - Mainz, Rhineland-Palatinate
  - Dresden, Saxony
  - Leipzig, Saxony
- Hungary (3):
  - Budapest
  - Debrecen
  - Pécs
- Italy (8):
  - Rome, Lazio
  - Genoa, Liguria
  - Milan, Lombardy
  - Turin, Piedmont
  - Cagliari, Sardinia
  - Sassari, Sardinia
  - Florence, Tuscany
  - Padua, Veneto
- Lithuania (2):
  - Kaunas
  - Vilnius
- Poland (8):
  - Bydgoszcz
  - Gdansk
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Poznan
  - Warsaw
- Portugal (5):
  - Coimbra
  - Leiria
  - Lisbon
  - Porto
  - Vila Franca de Xira
- Slovakia (4):
  - Bratislava
  - Nitra
  - Zvolen
  - Žilina
- Spain (5):
  - L'Hospitalet de Llobregat, Barcelona
  - San Cugat Del Vallès, Barcelona
  - Albacete
  - Barcelona
  - Valencia
- Switzerland (2):
  - Bern
  - Geneva
- United Kingdom (7):
  - Southampton, Hampshire
  - Camberley, Surrey
  - Guildford, Surrey
  - Newcastle upon Tyne, Tyne and Wear
  - Sunderland, Tyne and Wear
  - Leeds, West Yorkshire
  - London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at multiple study centers in 14 countries, between 19 November 2015 (first participant first visit) and 09 August 2017 (last participant last visit).
Pre-assignment Details: Overall, 676 participants were screened. Of them, 116 participants did not complete screening: 100 failed screening; 8 withdrew, 1 had an adverse event, 1 was lost to follow-up and 6 were not assigned to treatment for other reasons. A total of 560 participants were assigned to treatment and 31 participants discontinued the study prematurely.
Groups:
- Aflibercept: Participants were treated according to the EU-PI for treatment of DME for the first year of treatment and received 1 dose of 2 mg aflibercept injected IVT every 4 weeks for 5 consecutive doses, followed by dosing every 8 weeks thereafter until the end of the 52 week treatment period.
Period: Overall Study
Arm/Group | Aflibercept
Started | 560
Treated | 560
Completed | 529
Not Completed | 31
Not completed — Unspecified other | 3
Not completed — Adverse Event | 6
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by participant | 12
Not completed — Physician Decision | 1
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF) included all participants who received at least 1 injection of study drug.
Arm/Group | Aflibercept
Number analyzed (Participants) | 560
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Safety analysis set (SAF) included all participants who received at least 1 injection of study drug.
  years | 64.3 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: SAF included all participants who received at least 1 injection of study drug.
  Participants
    Female | 224
    Male | 336
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: SAF included all participants who received at least 1 injection of study drug.
  Participants
    American Indian or Alaska Native | 0
    Asian | 4
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 3
    White | 519
    More than one race | 0
    Unknown or Not Reported | 34
Central Retinal Thickness (CRT) [Mean (Standard Deviation); unit: microns] — The CRT was recorded at the study eye only. Participants received active treatment (intravitreal aflibercept) for the study eye and received close medical supervision. Population: FAS included all participants who received at least one injection of study drug and completed the baseline and at least one post-baseline NEI VFQ-25 questionnaire.
  microns
    number analyzed (Participants) | 553
    (all) | 465.08 (136.75)
Best Corrected Visual Acuity (BCVA) [Mean (Standard Deviation); unit: score on a scale] — The BCVA was recorded at the study eye only. Participants received active treatment (intravitreal aflibercept) for the study eye and received close medical supervision. Visual function was assessed using the ETDRS protocol (Early Treatment Diabetic Retinopathy Study Research Group 1985) starting at 4 meters. The values might range from 0 to 100. A higher score represents better functioning. Population: FAS included all participants who received at least one injection of study drug and completed the baseline and at least one post-baseline NEI VFQ-25 questionnaire.
  score on a scale
    number analyzed (Participants) | 553
    (all) | 61.5 (11.0)
NEI VFQ-25 total score [Mean (Standard Deviation); unit: score on a scale] — The NEI VFQ-25 consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. All items are scored so that a high score represents better functioning. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points, respectively. In this format scores represent the achieved percentage of the total possible score, example: a score of 50 represents 50% of the highest possible score. Population: FAS included all participants who received at least one injection of study drug and completed the baseline and at least one post-baseline national eye institute visual function questionnaire-25 (NEI VFQ-25) questionnaire.
  score on a scale
    number analyzed (Participants) | 553
    (all) | 70.224 (19.221)
NEI VFQ-25 near activities subscale [Mean (Standard Deviation); unit: score on a scale] — The NEI VFQ-25 near activities subscale was scored from 0-100 with a score of 0 being the worst outcome and 100 being the best outcome. Near activities are defined activities requiring near vision such as reading ordinary print in newspapers, performing work or hobbies requiring near vision, or finding something on a crowded shelf. Population: FAS included all participants who received at least one injection of study drug and completed the baseline and at least one post-baseline NEI VFQ-25 questionnaire.
  score on a scale
    number analyzed (Participants) | 553
    (all) | 62.967 (23.479)
NEI VFQ-25 distant activities subscale [Mean (Standard Deviation); unit: score on a scale] — The NEI VFQ-25 distant activities subscale was scored from 0-100 with a score of 0 being the worst outcome and 100 being the best outcome. Distant activities are defined as activities requiring distance vision, such as recognizing faces or reading street signs. Population: FAS included all participants who received at least one injection of study drug and completed the baseline and at least one post-baseline NEI VFQ-25 questionnaire.
  score on a scale
    number analyzed (Participants) | 553
    (all) | 71.964 (23.973)
Number of Participants with Diabetic Retinopathy Severity Score (DRSS) [Count of Participants; unit: Participants] — The following severities are possible. 10 = Diabetic retinopathy (DR) absent, 14 = DR questionable, 15 = DR questionable, 20 = Microaneurysms only, 35 = Mild Non-proliferative diabetic retinopathy (NPDR), 43 = Moderate NPDR, 47 = Moderately severe NPDR, 53 = Severe NPDR, 61 = Mild Proliferative diabetic retinopathy (PDR), 65 = Moderate PDR, 71 = High-risk PDR, 75 = High-risk PDR, 81 = Advanced PDR: fundus partially obscured, center of macula attached, 85 = Advanced PDR: posterior fundus obscured, or center of macula detached, 90 = cannot grade, even sufficiently for level 81 or 85. Population: FAS included all participants who received at least one injection of study drug and completed the baseline and at least one post-baseline NEI VFQ-25 questionnaire.
  Participants
    10 - DR absent: number analyzed (Participants) | 553
    10 - DR absent | 0
    15 - DR questionable: number analyzed (Participants) | 553
    15 - DR questionable | 2
    35 - Mild NPDR: number analyzed (Participants) | 553
    35 - Mild NPDR | 144
    43 - Moderate NPDR: number analyzed (Participants) | 553
    43 - Moderate NPDR | 184
    47 - Moderately severe NPDR: number analyzed (Participants) | 553
    47 - Moderately severe NPDR | 151
    53 - Severe NPDR: number analyzed (Participants) | 553
    53 - Severe NPDR | 48
    61 - Mild PDR: number analyzed (Participants) | 553
    61 - Mild PDR | 8
    65 - Moderate PDR: number analyzed (Participants) | 553
    65 - Moderate PDR | 8
    71 - High-risk PDR: number analyzed (Participants) | 553
    71 - High-risk PDR | 2
    90 - Cannot grade: number analyzed (Participants) | 553
    90 - Cannot grade | 6
Pre-injection Intraocular Pressure [Mean (Standard Deviation); unit: millimeter of mercury (mmHg)] — Population: SAF included all participants who received at least 1 injection of study drug.
  millimeter of mercury (mmHg) | 16.2 (3.0)
Systolic Blood Pressure [Mean (Standard Deviation); unit: millimeter of mercury (mmHg)] — Population: SAF included all participants who received at least 1 injection of study drug.
  millimeter of mercury (mmHg) | 138.1 (13.6)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: millimeter of mercury (mmHg)] — Population: SAF included all participants who received at least 1 injection of study drug.
  millimeter of mercury (mmHg) | 77.7 (9.4)
Heart Rate [Mean (Standard Deviation); unit: beats per minute (beats/min)] — Population: SAF included all participants who received at least 1 injection of study drug.
  beats per minute (beats/min) | 75.1 (10.1)
Body Temperature [Mean (Standard Deviation); unit: celsius] — Population: SAF included all participants who received at least 1 injection of study drug.
  celsius | 36.37 (0.38)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 52 in NEI VFQ-25 Total Score
Description: National eye institute 25-item visual function questionnaire (NEI VFQ-25) is a condition-specific measure which was designed to capture the specific impact of vision loss on health-related quality of life (HRQoL). The calculation for NEI VFQ-25 sub-scale scores and total score was performed according to the "NEI VFQ-25 Scoring Algorithm - August 2000". The NEI VFQ-25 consists of a base set of 25 vision-targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question. All items are scored so that a high score represents better functioning. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points, respectively. In this format scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score.
Time Frame: Baseline, Week 52
Population: FAS included all participants who received at least one injection of study drug and completed the baseline and at least one post-baseline NEI VFQ-25 questionnaire.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aflibercept
Number analyzed (Participants) | 553
score on a scale | 6.106 [5.303 to 6.909]

2. Secondary Outcome: Change From Baseline to Week 52 in the NEI VFQ 25 Near Activities Subscale
Description: NEI VFQ-25 is a condition-specific measure which was designed to capture the specific impact of vision loss on HRQoL. The calculation for NEI VFQ-25 sub-scale scores and total score was performed according to the "NEI VFQ-25 Scoring Algorithm - August 2000". Items within each sub-scale are averaged together to create the 12 sub-scale Scores. Items that are left blank (missing data) are not taken into account when calculating the scale scores. Sub-scales with at least one item answered can be used to generate a sub-scale score. Hence, scores represent the average for all items in the subscale that the respondent answered.The NEI VFQ-25 near activities subscale was scored from 0-100 with a score of 0 being the worst outcome and 100 being the best outcome. Near activities are defined as reading ordinary print in newspapers, performing work or hobbies requiring near vision, or finding something on a crowded shelf.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aflibercept
Number analyzed (Participants) | 553
score on a scale | 11.370 [10.108 to 12.632]

3. Secondary Outcome: Change From Baseline to Week 52 in the NEI VFQ 25 Distant Activities Subscale
Description: NEI VFQ-25 is a condition-specific measure which was designed to capture the specific impact of vision loss on HRQoL. The calculation for NEI VFQ-25 sub-scale scores and total score was performed according to the "NEI VFQ-25 Scoring Algorithm - August 2000". Items within each sub-scale are averaged together to create the 12 sub-scale Scores. Items that are left blank (missing data) are not taken into account when calculating the scale scores. Sub-scales with at least one item answered can be used to generate a sub-scale score. Hence, scores represent the average for all items in the subscale that the respondent answered. The NEI VFQ-25 distant activities subscale was scored from 0-100 with a score of 0 being the worst outcome and 100 being the best outcome. Distant activities are defined as activities requiring distance vision, such as recognizing faces or reading street signs.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aflibercept
Number analyzed (Participants) | 553
score on a scale | 7.331 [6.118 to 8.545]

4. Secondary Outcome: Change From Baseline to Week 52 in Best Corrected Visual Acuity (BCVA) (Early Treatment Diabetic Retinopathy Study [ETDRS] Letter Score])
Description: Visual function was assessed using the ETDRS protocol (Early Treatment Diabetic Retinopathy Study Research Group 1985) starting at 4 meters. The values might range from 0 to 100. A higher score represents better functioning.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aflibercept
Number analyzed (Participants) | 553
score on a scale | 10.0 [9.5 to 10.6]

5. Secondary Outcome: Change From Baseline to Week 52 in Central Retinal Thickness (CRT) Measured by Optical Coherence Tomography (OCT)
Description: Retinal and lesion characteristics were evaluated using spectral domain optical coherence tomography (OCT). For all visits where the OCT procedure was scheduled, images were captured and read by the investigator. All OCTs were electronically archived at the study sites as part of the source documentation.
Time Frame: Baseline, Week 52
Population: FAS included all participants who received at least one injection of study drug and completed the baseline and at least one post-baseline NEI VFQ-25 questionnaire. Participants who were evaluable for this measure at given time point for the arm were included in the category.
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | Aflibercept
Number analyzed (Participants) | 553
microns | -175.38 [-184.93 to -165.82]

6. Secondary Outcome: Proportion of Participants Progressing to Greater or Equal to (>=) 61 on the ETDRS Diabetic Retinopathy Severity Scale (DRSS) as Assessed by Fundus Photography (FP)
Description: The ETDRS DRSS was assessed by FP according to the following scale for both eyes. The following severities are possible.
  10 = Diabetic retinopathy (DR) absent, 14 = DR questionable, 15 = DR questionable, 20 = Micro-aneurysms only, 35 = Mild Non-proliferative diabetic retinopathy (NPDR), 43 = Moderate NPDR, 47 = Moderately severe NPDR, 53 = Severe NPDR, 61 = Mild Proliferative diabetic retinopathy (PDR), 65 = Moderate PDR, 71 = High-risk PDR, 75 = High-risk PDR, 81 = Advanced PDR: fundus partially obscured, center of macula attached, 85 = Advanced PDR: posterior fundus obscured, or center of macula detached, 90 = cannot grade, even sufficiently for level 81 or 85.
Time Frame: Baseline, Week 52
Population: Subjects in the FAS with gradable baseline and Week 52 FP and a DRSS of less than (<) 61 at baseline. Participants who were evaluable for this measure at given time point for the arm were included in the category.
Measure: Number; unit: proportion of participants
Arm/Group | Aflibercept
Number analyzed (Participants) | 553
proportion of participants | 0.4

7. Other Pre Specified Outcome: Change From Baseline in Pre-injection Intraocular Pressure for Study Eye Every 4 Weeks
Description: Intraocular pressure (IOP) was measured using applanation tonometry Goldmann, Tonopen or approved alternative). The same method of intraocular pressure measurement was used in each participant throughout the study. For the measurement of intraocular pressure, a local anesthetic combined with fluorescein was applied topically to the eye being tested (example: one drop of oxybuprocain plus fluorescein). In the below table, pre-injection intraocular pressure for study eye was reported.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 24, 32, 40, 48, 52
Population: SAF included all participants who received at least 1 injection of study drug. Participants who were evaluable for this measure at given time points for the arm were included in the categories.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Aflibercept
Number analyzed (Participants) | 560
millimeter of mercury (mmHg)
  Change at Week 4: number analyzed (Participants) | 552
  Change at Week 4 | -0.4 (2.9)
  Change at Week 8: number analyzed (Participants) | 545
  Change at Week 8 | -0.3 (2.9)
  Change at Week 12: number analyzed (Participants) | 547
  Change at Week 12 | -0.5 (2.9)
  Change at Week 16: number analyzed (Participants) | 548
  Change at Week 16 | -0.3 (2.9)
  Change at Week 24: number analyzed (Participants) | 542
  Change at Week 24 | -0.2 (3.0)
  Change at Week 32: number analyzed (Participants) | 541
  Change at Week 32 | -0.1 (3.0)
  Change at Week 40: number analyzed (Participants) | 533
  Change at Week 40 | 0.0 (3.0)
  Change at Week 48: number analyzed (Participants) | 532
  Change at Week 48 | 0.0 (3.0)
  Change at Week 52: number analyzed (Participants) | 527
  Change at Week 52 | 0.1 (3.1)

8. Other Pre Specified Outcome: Change From Baseline in Systolic Blood Pressure at Week 52
Description: Systolic blood pressure was measured in a consistent and standardized way according to locally established practice.
Time Frame: Baseline, Week 52
Population: SAF included all participants who received at least 1 injection of study drug. Participants who were evaluable for this measure at given time point for the arm were included in the category.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Aflibercept
Number analyzed (Participants) | 560
millimeter of mercury (mmHg) | -0.1 (15.1)

9. Other Pre Specified Outcome: Change From Baseline in Diastolic Blood Pressure at Week 52
Description: Diastolic blood pressure was measured in a consistent and standardized way according to locally established practice.
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Aflibercept
Number analyzed (Participants) | 560
millimeter of mercury (mmHg) | -0.3 (9.9)

10. Other Pre Specified Outcome: Change From Baseline in Heart Rate at Week 52
Description: Heart rate was measured in a consistent and standardized way according to locally established practice.
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: beats per minute (beats/min)
Arm/Group | Aflibercept
Number analyzed (Participants) | 560
beats per minute (beats/min) | -1.0 (9.5)

11. Other Pre Specified Outcome: Change From Baseline in Body Temperature at Week 52
Description: Temperature was measured in a consistent and standardized way according to locally established practice.
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: celsius
Arm/Group | Aflibercept
Number analyzed (Participants) | 560
celsius | -0.04 (0.41)

ADVERSE EVENTS:
Time Frame: From start of study treatment up to 30 days after the last injection of study treatment, up to week 52
Arm/Group | Aflibercept
All-Cause Mortality (participants affected / at risk) | 5/560
Serious Adverse Events (participants affected / at risk) | 66/560
Other Adverse Events (participants affected / at risk) | 0/560
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aflibercept (N=560)
Atrioventricular block (Cardiac disorders) | 1 (1)
Bundle branch block right (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 2 (3)
Cardiac failure chronic (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Anterior chamber inflammation (Eye disorders) | 1 (1)
Cataract subcapsular (Eye disorders) | 1 (1)
Posterior capsule opacification (Eye disorders) | 2 (2)
Vitreous haemorrhage (Eye disorders) | 1 (1)
Vitritis (Eye disorders) | 2 (2)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1)
Boutonneuse fever (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Diabetic foot infection (Infections and infestations) | 2 (2)
Endophthalmitis (Infections and infestations) | 3 (3)
Erysipelas (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Parotitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6)
Pyelonephritis chronic (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Inflammation of wound (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2)
Echocardiogram abnormal (Investigations) | 1 (1)
Influenza A virus test positive (Investigations) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3)
Lacunar stroke (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Vascular encephalopathy (Nervous system disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Major depression (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 2 (2)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Umbilical hernia repair (Surgical and medical procedures) | 1 (1)
Vitrectomy (Surgical and medical procedures) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2)
Peripheral vascular disorder (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Center provides publication/presentation related to the Study Drug/Results 60 days prior to due date submission/presentation allowing Bayer review. Center receives notification within 45 days, Center reminds Bayer of Publication´s due date. Expected comments are within 60 days, if not Center to publish. Multi-center´s Results publication coordinates through Bayer Center publishes their Results provided overall results haven't been published within 18 months from Study completion for compliance.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-05-04): https://cdn.clinicaltrials.gov/large-docs/95/NCT02581995/SAP_000.pdf
  • Study Protocol (2015-09-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT02581995/Prot_001.pdf